CLINICAL TRIAL: NCT03366376
Title: A Phase II Multi-institutional Study of Hippocampus-sparing Whole Brain Radiotherapy and Simultaneous Integrated Boost for Multiple Brain Metastases From Non-small Cell Lung Cancer
Brief Title: Hippocampus-sparing WBRT and Simultaneous Integrated Boost for Multiple Brain Metastases From NSCLC
Acronym: KROG17-06
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Korean Radiation Oncology Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-08-070
Record Dates: First submitted 2017-12-03; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Brain Metastases
Keywords: hippocampus; radiotherapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): WBRT with hippocampus-sparing and SIB
  Interventions: Radiation: WBRT with hippocampus-sparing and SIB

INTERVENTIONS:
Radiation: WBRT with hippocampus-sparing and SIB — Radiotherapy could be delivered in 5, 8, or 10 fractions according to participating investigator's choice. The prescribed doses are as below;
  Fractions 5fxs 8fxs 10fxs Whole brain 20 Gy 24 Gy 25 Gy Gross tumor 30 Gy 40 Gy 40 Gy

SUMMARY:
This study evaluates hippocampus-sparing whole-brain radiotherapy with simultaneous integrated boost for patients with multiple brain metastases from non-small cell lung cancer. The primary endpoint is intracranial progression free survival, and secondary endpoints are verbal neurocognitive function, overall survival, adverse events according to CTCAE v4.03, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of primary non-small cell lung cancer
* 3 or more measurable brain metastasis ≥3 mm outside a 5-mm margin around either hippocampus on gadolinium contrast enhanced MRI within 14 days prior to registration
* KPS ≥70
* Age ≥55 years
* Informed consent prior to study entry

Exclusion Criteria:

* Patients with leptomeningeal metastases
* ≥3 organ sites of extracranial metastases (including lung-to-lung metastases) within 3 months
* Contraindication to MRI such as implanted metal devices or foreign bodies
* Prior radiation therapy (including SRS) to the brain

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-12-11 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression free survival | until 12 months
  Time from the date of start of radiotherapy to the date of death or intracranial progression

SECONDARY OUTCOMES:
Verbal neurocognitive function (Seoul Verbal Learning Test-Elderly, SVLT-E) | 3,6,12 months
  The relative decline in SVLT-E score from baseline to below time frame; ΔSVLT = (SVLTB - SVLTF) ÷ SVLTB, where B=baseline and F=follow-up.
Overall survival | until 12 months
  Time from the date of start of radiotherapy to the date of death from any cause
Adverse events | 3,6,12 months
  CTCAE v4.03
Quality of life | 3,6,12 months
  EORTC QLQ-C30 and BN20

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No